CLINICAL TRIAL: NCT02234648
Title: Investigate the Effect of Tart Montmorency Cherry Juice (Prunus Cerasus) on Vascular Function.
Brief Title: To Investigate the Effect of Tart Montmorency Cherry Juice (Prunus Cerasus) on Vascular Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Glyn Howatson, Dr., Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NUKK1
Record Dates: First submitted 2014-09-01; First posted 2014-09-09 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: Vascular Function; tart Montmorency cherries; Arterial Stiffness; Blood Flow
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The PLA supplement consisted of a commercially available, less than 5% fruit, cordial (Protein - Trace, Carbohydrate 260 mg•mL-1, Sodium 0.02 mg•mL-1, Fibre-Trace and Anthocyanins-Trace for colour), mixed with water, whey protein isolate (Arla Foods Ltd., Leeds, UK) and maltodextrin (MyProtein Ltd., Northwich, UK) until matched for carbohydrate and calorie content of the MC.
  Interventions: Other: Placebo
- 60mL tart Montmorency cherry juice (Active Comparator): One bolus of 60mL of tart Montmorency cherry (MC) juice mixed with 100mL of water. Independent analysis of MC (Atlas Biosciences, 2010) provided the following compositional data; Fat 0.028 mg•mL-1, Protein 31.47 mg•mL-1, Carbohydrate 669.4 mg•mL-1, Cholesterol < 0.01 mg•mL-1, Sodium 0.691 mg•mL-1, Calcium 0.137 mg•mL-1 and Iron 0.026 mg•mL-1. Additionally, according to the manufacturers guidelines (Cherry Active, Hanworth, UK),
  Interventions: Dietary Supplement: 60mL tart Montmorency cherry juice

INTERVENTIONS:
Dietary Supplement: 60mL tart Montmorency cherry juice — One bolus of 60mL of tart Montmorency concentrate mixed with 100mL of water.
  Arms: 60mL tart Montmorency cherry juice
Other: Placebo — One bolus of less than 5% fruit cordial mixed with water, maltodextrin and whey protein isolate to match for carbohydrate and calorie content of the juice.
  Other Names: less than 5% "Kia Ora" mixed fruit squash
  Arms: Placebo

SUMMARY:
Given the global health issues associated with poor cardiovascular function, interventions that help reduce the severity, with emphasis on prevention would not only have economic implications, but would also improve health, wellbeing and quality of life. Research provides evidence that consumption of a diet high in plant foods and rich is polyphenols is associated with a reduction in the incidence of cardiovascular disease (Hung et al 2004). Tart Montmorency cherries have been shown to be high in numerous phytochemicals (Wang et al 1999; Seeram et al 2001). Several of these compounds, are known to be vasoactive and improve blood vessel function by increasing bioavailability of vasodilators (Mudnic et al 2012), reducing vasoconstrictors (Broncel et al 2010), decreasing platelet aggregation (Hubbart et al 2006) and increasing blood vessel dilation (Schroeter et al 2006). Impaired function of the lining of blood vessels (endothelial dysfunction) has been linked to increased risk of cardiovascular disease. However, the bioavailability of all the compounds in Tart Montmorency Cherry Juice and their efficacy with respect to vascular function has not been fully determined. This study will examine the influence of tart Montmorency cherry juice on cardiovascular function, specifically arterial stiffness by pulse wave velocity and blood flow in the microcirculation by laser Doppler imaging. This study will also examine digital volume pulse and pulse wave analysis. These data will provide information on the ability of TMCJ to affect blood flow and vascular function.

DETAILED DESCRIPTION:
Participants provided blood samples immediately before supplementation and sequentially 8h post ingestion. Additionally, vascular measurements including laser Doppler imaging (LDI), pulse wave analysis (PWA), pulse wave velocity (PWV), digital volume pulse (DVP) and blood pressure (BP) were performed with the participant in a supine position. LDI, PWV, PWA, and DVP were measured at 1, 2, 3, 5 and 8h intervals. BP was performed at hourly intervals. All vascular measurements took place on the non - cannulated arm. No additional food or fluid was provided during the study period except for low-nitrate mineral water. Following a minimum of two weeks washout, the participants were required to return to the laboratory to repeat the procedure with the other intervention drink.

ELIGIBILITY:
Inclusion Criteria:

* Those with blood pressure below 140/90
* Males
* Aged 21 - 55y

Exclusion Criteria:

* Those with blood pressure above 140/90
* Taken other medication/ supplements.
* Those aged >21 or <55.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in microvasculature blood flow | 0,1,2,3,5 and 8 hours

SECONDARY OUTCOMES:
Changes in arterial stiffness | 0,1,2,3,5 and 8 hours
Changes in blood pressure | 0,1,2,3,4,5,6,7 and 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (2):
- United Kingdom (2):
  - Northumbria University, Newcastle upon Tyne, Newcastle Upon Tyne
  - Northumbria University, Newcastle upon Tyne

REFERENCES:
- [Derived] Keane KM, George TW, Constantinou CL, Brown MA, Clifford T, Howatson G. Effects of Montmorency tart cherry (Prunus Cerasus L.) consumption on vascular function in men with early hypertension. Am J Clin Nutr. 2016 Jun;103(6):1531-9. doi: 10.3945/ajcn.115.123869. Epub 2016 May 4. PMID 27146650